CLINICAL TRIAL: NCT01401907
Title: Randomized Study of Early Palliative Care Integrated With Standard Oncology Care Versus Standard Oncology Care Alone in Patients With Advanced Lung and Non-colorectal Gastrointestinal Malignancies
Brief Title: Early Palliative Care in Advanced Lung and Gastrointestinal Malignancies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Jennifer Temel, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 10-434
Record Dates: First submitted 2011-07-20; First posted 2011-07-25 (Estimated); Results first posted 2017-07-13 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Non-small Cell Lung Cancer; Small Cell Lung Cancer; Mesothelioma; Esophageal Cancer; Gastric Cancer; Liver Cancer; Pancreatic Cancer
Keywords: Palliative care; Lung; Gastric; Liver; Pancreatic; Esophageal; Caregiver
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma; Mesothelioma; Esophageal Neoplasms; Stomach Neoplasms; Liver Neoplasms; Pancreatic Neoplasms

STUDY DESIGN:
Intervention Model Description: early palliative care
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Early Palliative Care (Experimental): Subjects receive standard of care with early palliative care.
  Interventions: Other: early palliative care
- Standard of Care (No Intervention): Subjects receives standard of care

INTERVENTIONS:
Other: early palliative care — patient assigned to the intervention will receive early palliative care along with standard oncology care.
  Arms: Early Palliative Care

SUMMARY:
The purpose of this study is to compare two types of care - standard oncology care and standard oncology care with early palliative care (started soon after diagnosis) to see which is better for improving the experience of patients and families with advanced lung and non-colorectal GI cancer. The study will use questionnaires to measure patients' and caregivers' quality of life, mood, coping and understanding of their illness.

DETAILED DESCRIPTION:
Subjects and their caregiver will complete a baseline questionnaire and then be randomized to a study group.

Subjects who are randomized to Standard Oncology Care will follow up with their treating oncologist. They will consult with the palliative care team at their request or at the request of the treating oncologist. They will complete questionnaires at 12 weeks and 24 weeks after enrollment.

Subjects who are randomized to the Standard Oncology Care with Early Palliative Care will meet with a palliative care clinician at their next medical oncology visit or infusion visit. They will meet with the palliative care clinician at least every three weeks. They will complete questionnaires at 12 and 24 weeks after enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed metastatic lung cancer (NSCLC, small cell lung cancer, and mesothelioma)or non-colorectal GI cancer (esophageal, gastric and hepatobiliary) not being treated with curative intent
* Informed of metastatic disease within the previous 8 weeks
* No prior therapy for metastatic disease
* Able to read questions in English or willing to complete questionnaires with the assistance of an interpreter
* Relative or friend of patient who will likely accompany the patient to clinic visits

Exclusion Criteria:

* Significant psychiatric or other co-morbid disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 351 (Actual)
Dates: Start 2011-05; Primary Completion 2016-04 (Actual); Study Completion 2019-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Temel, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
will share deidentified data with proper IRB approval

REFERENCES:
- [Derived] Hoerger M, Greer JA, Jackson VA, Park ER, Pirl WF, El-Jawahri A, Gallagher ER, Hagan T, Jacobsen J, Perry LM, Temel JS. Defining the Elements of Early Palliative Care That Are Associated With Patient-Reported Outcomes and the Delivery of End-of-Life Care. J Clin Oncol. 2018 Apr 10;36(11):1096-1102. doi: 10.1200/JCO.2017.75.6676. Epub 2018 Feb 23. PMID 29474102
- [Derived] Greer JA, Jacobs JM, El-Jawahri A, Nipp RD, Gallagher ER, Pirl WF, Park ER, Muzikansky A, Jacobsen JC, Jackson VA, Temel JS. Role of Patient Coping Strategies in Understanding the Effects of Early Palliative Care on Quality of Life and Mood. J Clin Oncol. 2018 Jan 1;36(1):53-60. doi: 10.1200/JCO.2017.73.7221. Epub 2017 Nov 15. PMID 29140772

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Early Palliative Care | Standard of Care
Started | 175 | 175
12 Week Outcomes | 148 | 153
Completed (24 week outcomes) | 118 | 124
Not Completed | 57 | 51

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Early Palliative Care | Standard of Care | Total
Number analyzed (Participants) | 175 | 175 | 350
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.64 (11.26) | 64.03 (10.46) | 64.85 (10.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 84 | 77 | 161
  Male | 91 | 98 | 189
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 2 | 9
  Not Hispanic or Latino | 168 | 173 | 341
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 0 | 4
  Asian | 5 | 3 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 4 | 10
  White | 156 | 167 | 323
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Functional Assessment of Cancer Therapy (Quality of Life Measure)
Description: The Functional Assessment of Cancer Therapy - General is a quality of life measure with higher scores indicating better quality of life (range 0-108). We are examining the adjusted mean difference from baseline to 12 weeks in this study
Time Frame: 12 weeks
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Early Palliative Care | Standard of Care
Number analyzed (Participants) | 148 | 153
units on a scale | 81.10 [78.11 to 82.08] | 77.70 [75.77 to 79.63]

2. Secondary Outcome: Functional Assessment of Cancer Therapy (Quality of Life Measure)
Description: The Functional Assessment of Cancer Therapy - General is a quality of life measure with higher scores indicating better quality of life (range 0-108). We are examining the adjusted mean difference from baseline to 24 weeks.
Time Frame: 24 weeks
Population: The analysis focuses on participants who completed week-24 questionnaires (N = 118 in the early palliative care arm, and N = 124 in the standard of care arm)
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Early Palliative Care | Standard of Care
Number analyzed (Participants) | 118 | 124
units on a scale | 81.26 [78.89 to 83.63] | 75.90 [73.59 to 78.21]

3. Secondary Outcome: Rate of Clinically Significant Depression Symptoms Based on Hospital Anxiety and Depression Scale
Description: The hospital anxiety and depression scale examines symptoms of depression and anxiety. We compared rates of clinically significant depression symptoms (using a cut off of 8 on the depression subscale score) between study arms at week-12 and week-24.
Time Frame: Week-12 and Week-24
Population: The two rows examine outcomes at two different time points week-12 and week-24. Please note the number of participants included in week-12 and week-24 analyses reflect the participants who completed the hospital anxiety and depression scale at these time points (study completers), which explains the discrepancy with the flow chart.
Measure: Count of Participants; unit: Participants
Arm/Group | Early Palliative Care | Standard Oncology Care
Number analyzed (Participants) | 138 | 141
Participants
  Week-12 | 29 | 32
  Week-24: number analyzed (Participants) | 118 | 122
  Week-24 | 24 | 32

4. Secondary Outcome: Number and Percentage of Participants Who Reported Goal of Their Cancer Treatment is to Cure Their Cancer
Description: We used the response to an item on Perception of Treatment and Prognosis Questionnaire to compare rates of accurate prognostic understanding between study arms. Participants reported their primary goal of their current cancer treatment: 1) to cure my cancer; 2) to lesson my suffering as much as possible; 3) for me and/or my family to be able to keep hoping; 4) to make sure I have done everything; 5) to extend my life as long as possible; 6) to help cancer research. Participants' responses were dichotomized as 1) to cure my cancer vs. all other.
Time Frame: Week12 and Week 24
Population: The different rows reflect analyses at week-12 and week-24. Please note the number of participants included in week-12 and week-24 analyses reflect the participants who completed the Perception of Treatment and Prognosis Questionnaire at these time points (study completers), which explains the discrepancy with the flow chart.
Measure: Count of Participants; unit: Participants
Arm/Group | Early Palliative Care | Standard Oncology Care
Number analyzed (Participants) | 143 | 145
Participants
  Goal Cure Week-12 | 41 | 50
  Goal Cure Week-24: number analyzed (Participants) | 115 | 116
  Goal Cure Week-24 | 37 | 32

5. Secondary Outcome: Family Caregiver Quality of Life as Measured by the SF-36
Description: The Medical Health Outcomes Survey- Short Form (SF-36) is a measure of QOL. The SF-36 measures eight domains of health-related quality of life: physical functioning, role limitation due to physical health, bodily pain, general health perceptions, vitality, social functioning, role limitation due to emotional health, and mental health. The response choices are scored and summed to yield two physical (PCS) and mental (MCS) component summary measures with ranges from 0-100. Higher scores indicate better quality of life. We compared family caregiver PCS and MCS scores between the two study arms at week-12 and week-24 adjusting for baseline scores.
Time Frame: Week-12 and Week-24
Population: Adjusted Means controlling for baseline scores. The different rows reflect Week-12 and Week-24 outcomes on SF-36 PCS and MCS domains. The number of participants included in week-12 and week-24 analyses reflect the participants who completed the SF-36 at these time points, which explains the discrepancy with the flow chart.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Early Palliative Care | Standard Oncology Care
Number analyzed (Participants) | 110 | 119
units on a scale
  SF36 PCS Week-12 | 52.94 [51.30 to 54.59] | 51.40 [49.83 to 52.98]
  SF36 MCS Week-12 | 47.00 [45.26 to 48.74] | 45.92 [44.25 to 47.59]
  SF36 PCS Week-24: number analyzed (Participants) | 89 | 94
  SF36 PCS Week-24 | 52.71 [51.02 to 54.40] | 53.22 [51.58 to 54.86]
  SF36 MCS Week-24: number analyzed (Participants) | 89 | 94
  SF36 MCS Week-24 | 46.21 [44.09 to 48.33] | 45.59 [44.09 to 48.33]

6. Secondary Outcome: Family Caregiver Psychological Distress (Based on the Hospital Anxiety and Depression Scale)
Description: We used the Hospital Anxiety and Depression scale to measure overall psychological distress in family caregivers. The Hospital Anxiety and Depression Scale contains two subscales measuring depression and anxiety respectively. When examined continuously, this scale reflects degree of psychological distress with higher scores indicating more psychological distress (range 0-42). We compared overall psychological distress (HADS-total) among family caregivers between the two study arms
Time Frame: Week 12 and Week 24
Population: Looking at the HADS-total score at week-12 and week-24. Please note the number of participants included in week-12 and week-24 analyses reflect the participants who completed the hospital anxiety and depression scale at these time points (study completers), which explains the discrepancy with the flow chart.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Early Palliative Care | Standard Oncology Care
Number analyzed (Participants) | 110 | 119
units on a scale
  HADS-Total Week-12 | 9.02 [8.09 to 9.96] | 10.48 [9.58 to 11.38]
  HADS-Total Week-24: number analyzed (Participants) | 89 | 94
  HADS-Total Week-24 | 9.82 [8.65 to 10.99] | 10.72 [8.65 to 10.99]

7. Secondary Outcome: Number and Percentage of Family Caregivers Who Reported the Goal of Treatment is to Cure Cancer
Description: We used the response to an item on Perception of Treatment and Prognosis Questionnaire to compare rates of accurate prognostic understanding between study arms. Family caregivers reported their primary goal of the current cancer treatment: 1) to cure my cancer; 2) to lesson my suffering as much as possible; 3) for me and/or my family to be able to keep hoping; 4) to make sure I have done everything; 5) to extend my life as long as possible; 6) to help cancer research. Family caregivers' responses were dichotomized as 1) to cure my cancer vs. all other.
Time Frame: 12 and 24 weeks
Population: Proportion of caregiver goal is cure at week-12 and week-24. Please note the number of participants reflect those who completed the Perception of Treatment and Prognosis Questionnaire at week-12 and week-24, which explains the discrepancy with the participants flow.
Measure: Count of Participants; unit: Participants
Arm/Group | Early Palliative Care | Standard Oncology Care
Number analyzed (Participants) | 106 | 113
Participants
  Goal Cure Week-12 | 34 | 40
  Goal Cure Week-24: number analyzed (Participants) | 85 | 89
  Goal Cure Week-24 | 19 | 29

8. Secondary Outcome: Coping (Brief Cope)
Description: compare mean change in approach oriented coping from baseline to week-24. Approach oriented coping scale is composed of active coping, positive reframing, and acceptance subscales. Scores range from 0-8 with higher scores indicate higher approach-oriented coping
Time Frame: Up to week-24
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Early Palliative Care | Standard Oncology Care
Number analyzed (Participants) | 118 | 124
units on a scale | 0.21 [-0.39 to 0.81] | -0.88 [-1.50 to -0.27]

ADVERSE EVENTS:
Time Frame: 6 months
Description: no AE from this non-medication/treatment study
Arm/Group | Early Palliative Care | Standard of Care
All-Cause Mortality (participants affected / at risk) | 27/175 | 32/175
Serious Adverse Events (participants affected / at risk) | 0/175 | 0/175
Other Adverse Events (participants affected / at risk) | 0/175 | 0/175

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No